CLINICAL TRIAL: NCT02307877
Title: Comparative Effectiveness of Long Term Fingolimod Versus Glatiramer Acetate on Brain Atrophy Rates, Cognition and Patient Reported Outcomes in Patients With Multiple Sclerosis
Brief Title: Comparison of Brain Atrophy Rates, Cognition, and Patient-Reported Outcomes in MS Patients Using Long-term Fingolimod and Glatiramer Acetate
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0774; UL1TR001082 (NIH)
Record Dates: First submitted 2014-08-26; First posted 2014-12-04 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fingolimod: Subjects currently taking Fingolimod for a minimum of 2 years
- glatiramer acetate: Subjects currently taking glatiramer acetate for a minimum of 2 years

SUMMARY:
Rates of brain atrophy for long term users of fingolimod when compared to glatiramer acetate have not been examined in patients with relapsing forms of multiple sclerosis (MS). As patients on long term therapy typically have little or no overt signs of white matter inflammatory activity (T2, gad lesions), brain atrophy measures can provide insight into whether there is continued progression of MS in these patients. What remains unknown is whether patients on a particular therapy have a slower rate of brain atrophy. This would provide convincing evidence that central nervous system tissue injury is further suppressed. Such information would be of substantial clinical benefit when deciding between various therapies.

The investigators will estimate the impact of long term use of fingolimod therapy (defined as a minimum of two years on therapy) on whole brain atrophy in treated patients with relapsing forms of MS as compared to age and gender matched patients on Glatiramer Acetate.

The investigators secondary goal is to determine the correlation between brain atrophy and cognitive performance in treated patients with relapsing forms of MS.

The investigators will also examine the correlation between the NeuroQualityofLife (NeuroQOL) PROs, patient self-reports of disability, clinical assessment of physical disability, work productivity, clinical assessments of cognitive functioning with whole brain volume loss for patients on long term fingolimod vs. long term glatiramer acetate therapy matched on age and gender.

The investigators anticipate the findings of this study will generate relevant hypotheses about these relationships.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent
* Between 18-55 years of age at the time of informed consent.
* Diagnosis of any form of MS as defined by the 2010 revised McDonald criteria
* Currently taking fingolimod or glatiramer acetate for a minimum of two years at the time of the initial baseline visit
* Must be willing and able to comply with the protocol requirements for the duration of the study

Exclusion Criteria:

* Suffering from comorbidities that could confound the MRI outcomes or are (relative) contraindicated to receive treatment with fingolimod such as:

  * diabetes,
  * myocardial infarction,
  * unstable angina,
  * transient ischemic attack,
  * decompensated heart failure,
  * history of Mobitz Type II 2nd or 3rd degree atrioventricular block,
  * sick sinus syndrome,
  * history of stroke,
  * history of traumatic brain injury,
  * history of encephalitis,
  * dementia (not related to MS).
* Systemic steroid used (oral or IV) within 30 days of the baseline visit.
* Ever treated with chemotherapy.
* Ever having undergone cranial radiation, or intracranial surgery.
* Unable to tolerate an MRI scan.
* Is pregnant or breastfeeding or planning on pregnancy during the study period.
* Is decisionally challenged, illiterate or blind
* Is non-English speaking (as the PRO instruments are only validated in English)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS patients who have been taking either fingolimod or glatiramer acetate for at least 2 years
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Whole Brain Atrophy (Rate of whole brain atrophy (T2 - T0): Two-time point percentage brain volume change (PBVC) | Baseline; Year 1; Year 2.
  Rate of whole brain atrophy (T2 - T0): Two-time point percentage brain volume change (PBVC) over the two years of the study will be estimated from the 3D T-1 weighted acquisition with Structural Image Evaluation Using Normalization of Atrophy (SIENA) software, part of FSL (Functional MRI of the Brain [FMRIB] Software Library, http://www.fmrib.ox.ac.uk/fsl).

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Nair, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States